CLINICAL TRIAL: NCT04754295
Title: Effect of Goal-directed Fluid Management Guided by Non-invasive Device on Incidence of Postoperative Complications in Neurosurgery: Pilot Study
Brief Title: Goal-directed Therapy in Neurosurgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ondrej Hrdy, Principal Investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT0012021
Record Dates: First submitted 2021-02-02; First posted 2021-02-15 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Surgery--Complications
Keywords: Neurosurgery; Goal-Directed Therapy; Complications; Pilot study
MeSH Terms: interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STANDARD (Experimental): In this arm standard monitoring of vital signs will be used during operation.
  Interventions: Other: STANDARD
- GDT (Experimental): A non-invasive hemodynamic monitor STARLINK™SV will be used in addition to standard monitoring.
  Interventions: Other: Goal-Directed Therapy

INTERVENTIONS:
Other: Goal-Directed Therapy — Administration of fluids and vasoactive drugs guided by non-invasive haemodynamic monitoring
  Arms: GDT
Other: STANDARD — Administration of fluids and vasoactive drugs guided by standard vital signs monitoring
  Arms: STANDARD

SUMMARY:
The purpose of the study is to assess feasibility of future large randomised controled study aimed on assessment of effect of goal-directed therapy on incidence of complications in neurosurgery compared to standard care.

DETAILED DESCRIPTION:
Patients undergoing neurosurgical operations are at risk of inadequate intravascular volume for several reasons. The appropriate fluid management in neurosurgery is a challenge. Goal-directed therapy has been shown to improve the outcome of patients undergoing major surgery. Current knowledge regarding effect of fluid management on patient-orientated outcomes in neurosurgery is limited.

This study is designed as a pilot study with two parallel groups. Patients scheduled to planned brain surgery at the University Hospital Brno will be screened whether they meet the inclusion criteria. After obtaining informed consent, the patient will be randomized to one of the study arms.

In one arm (STANDARD) standard monitoring of vital signs will be introduced. During the operation, perioperative fluid therapy and administration of vasoactive agents will depend entirely at the discretion of the attending anaesthetist. Postoperative therapy will be fully controlled and will depend on the decision of the attending physician. In the second arm (GDT), a non-invasive hemodynamic monitor STARLINK™SV will be introduced in addition to standard monitoring. In this arm, basal infusion with crystalloid balanced solution will be initiated. Additional boluses of fluids will be administered based on haemodynamic monitoring. The primary outcome of the study is a proportion of patients with serious adverse event (SAE). Incidence of SAEs will be compared between study groups. SAE will be defined as unsatisfactory brain tissue relaxation at the end of operation and any intervention for brain oedema postoperatively.

The secondary outcome is to compare proportion of patients with postoperative complications in both groups and length of ICU and hospital stay.

This study will enroll 34 patients in total, 17 in each group. After completion of enrolment of patients the statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* anticipated duration of surgery at least 2 hours
* signed written consent form
* American Society of Anesthesiologists (ASA) classification < 4.

Exclusion Criteria:

* unavailability of hemodynamic monitor
* emergency operation
* ASA ≥4
* sitting operating position and awake craniotomy
* awake craniotomy
* serious cardiorespiratory disorder
* cardiac arrythmia
* obesity with BMI above 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events 1 | During the Surgery
  Assessment of number of patients with serious adverse event (SAE). SAE is defined as unsatisfactory brain tissue relaxation at the end of surgery assessed by neurosurgeon. Level 3 or 4 of brain tissue relaxation will be considered as unsatisfactory (level 1 - completely relaxed, level 2 - satisfactorily relaxed, level 3 - firm, level 4 - bulging).
Serious Adverse Events 2 | 24 hours postoperatively
  Assessment of number of patients with serious adverse event (SAE). SAE is defined as any intervention indicated for treatment of brain edema 24 hours after surgery.
Recruitment rate | through study completion, an average of 6 months
  Proportion of eligible patients who consent to participate in the study.
Completeness of Case Report Forms | through study completion, an average of 6 months
  Proportion of enrolled patients with completed Case Report Form.

SECONDARY OUTCOMES:
Complications | through study completion, an average of 6 months
  Number of patients with pre-defined postoperative complication.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, M.D., Ph.D., Principal Investigator — Masaryk University Brno and University Hospital
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hrdy O, Duba M, Dolezelova A, Roskova I, Hlavaty M, Traj R, Bonisch V, Smrcka M, Gal R. Effects of goal-directed fluid management guided by a non-invasive device on the incidence of postoperative complications in neurosurgery: a pilot and feasibility randomized controlled trial. Perioper Med (Lond). 2023 Jul 5;12(1):32. doi: 10.1186/s13741-023-00321-3. PMID 37408018